CLINICAL TRIAL: NCT00128726
Title: The Effects of Continuous Administration of a Monophasic Oral Contraceptive on Bleeding Days and Endometrial and Ovarian Function
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Other Study IDs: HY01-190; R01HD043332 (NIH)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Menstrual Cycle; Healthy
Keywords: continuous combined oral contraceptive; endometrial and ovarian suppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urines, tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a continuous combined oral contraceptive pill (CCOCP) regimen. The investigators hypothesize that there will be a decrease in the number of vaginal bleeding days in the continuous regimen compared to a traditional 21/7 regimen. In addition, the investigators hypothesize that there will be increased endometrial and ovarian suppression in the CCOCP regimen.

DETAILED DESCRIPTION:
In the U.S. many women of reproductive age use some form of contraception, 23% of whom use estrogen-progesterone combined oral contraceptives. Low-dose oral contraceptives suppress ovulation and dominant follicle selection by inhibiting luteinizing hormone and follicle stimulating hormone secretion by the pituitary gland. Under social, cultural and religious influences, women have traditionally been prescribed oral contraceptives in a pattern of 21 days of active pills with seven days of inactive pills as a way of mimicking the natural menstrual cycle and provide reassurance of the absence of pregnancy by a withdrawal bleed during the placebo period. However, the withdrawal bleeding that occurs during the placebo period may still present with debilitating menstrual symptoms such as cramping, spotting break through bleeding, menstrual migraines and anemia. These menstrual disorders remain one of the most common reasons for prescribing the oral contraceptives. Suppression of bleeding by discarding the seven placebo tablets has been advocated for women with severe mental disabilities that impair hygiene and proper use, as well as for occasional use by women inconvenienced by menstruation (i.e. female athletes during competition and women in the military). Additionally, many physicians have used oral contraceptive pill regimens to treat endometriosis, premenstrual syndrome, anovulatory dysfunctional uterine bleeding, acne, hirsutism and anemia. The seven day pills free ovarian axis and ovarian follicular development and increase ovarian sex steroid production which may result in mild exacerbations of the treated condition. There is a growing patient preference to avoid vaginal bleeding completely, both in pre-menopausal and post-menopausal hormone replacement regimens in the general population. This is reflected in a woman's attitude about changing menstrual bleeding patterns as assessed by a 1996 Dutch survey. The majority of women in all studied age groups said that they would prefer decreasing the frequency of bleeding to less than once a month or completely eliminating menses altogether through the use of oral contraceptives. Therefore, reducing bleeding days is an important goal for improving quality of life in women suffering from the discomfort and inconvenience of withdrawal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of legal age of consent between 18-35 years who wish to use a continuous combined oral contraceptive and are non-smokers.
* Must have a regular (25-31) day menstrual cycle for the three month period preceding enrollment.
* Subject will comply with protocol, in the opinion of the investigator.

Exclusion Criteria:

* Thrombophlebitis
* Known or suspected clotting disorders
* Cerebrovascular or coronary artery disease or myocardial infarction
* Malignancy
* Known or suspected estrogen dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Benign or malignant liver tumor that developed during the use of oral contraceptives or other estrogen-containing products
* Hyperlipidemia - fasting cholesterol level greater than 6.73 mmol/L (260mg); fasting triglyceride level greater than 3.39 mmol/L (300mg/dl); high cholesterol.
* Diabetes mellitus
* Migraine or increased sensitivity of headaches during previous estrogen or oral contraceptive study
* Depression requiring hospitalization or associated with suicidal ideation
* Chronic renal disease
* Known hypersensitivity to estrogens and/or progestogens
* Neuro-ocular disorders
* Cholestatic jaundice
* Pregnancy while taking oral contraceptives
* Persistent non compliance with taking medication
* Serious adverse experiences with oral contraceptive use
* Malabsorption due to illness or surgery
* Use of any experimental drug or device within the last 90 days before study drug administration
* Any anticonvulsant medications
* Any use of rifampin within 3 months of enrollment
* Any use of lipid lowering agents
* Impaired liver function or disease
* Known or suspected pregnancy
* Hypertension whether treated or untreated
* Cervical cytological smear or low grade squamous intraepithelial lesion (SIL) or greater that is untreated within the last year
* The use of an intrauterine device (IUD) or injectable or implantable estrogen, progestogens, or androgens during the six month period before enrollment; or oral contraceptive or sex hormone use within three cycles before enrollment.
* Breast feeding
* Known or suspected alcoholism or drug abuse
* Smoking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women between 18-35 years of age who wish to use a continuous combined oral contraceptive and are non-smokers. Must have regular menstrual cycles for a 3 month period.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2001-06; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Principal Investigator — The Penn State Hershey Medical Center/College of Medicine
Locations (1):
- The Penn State Hershey Medical Center, Hershey, Pennsylvania, United States